CLINICAL TRIAL: NCT04040946
Title: Phase III Trial Comparing 2 Diagnostic Strategies for Preoperative Localization of Parathyroid Adenoma in Primary Hyperparathyroidism:TEMP / CT With Tc99m-sestaMIBI or PET / CT With F18-choline in First Intention
Brief Title: Trial Comparing 2 Diagnostic Strategies for Preoperative Localization of Parathyroid Adenoma in Primary Hyperparathyroidism:TEMP / CT With Tc99m-sestaMIBI or PET / CT With F18-choline in First Intention
Acronym: APACH2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APACH2
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Parathyroid Adenoma; Hyperparathyroidism; F18-choline
MeSH Terms: conditions — Parathyroid Neoplasms; Hyperparathyroidism

STUDY DESIGN:
Intervention Model Description: Open, randomized, phase III study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEMP-TDM with MIBI (Other): Performing a MIBI scintigraphy, then, in the case of negativity, a F18-choline PET
  Interventions: Diagnostic Test: MIBI scintigraphy; Diagnostic Test: F18-choline PET
- F18-choline PET (Other): Realization of F18-choline PET, then, in case of negativity, a MIBI scintigraphy
  Interventions: Diagnostic Test: MIBI scintigraphy; Diagnostic Test: F18-choline PET

INTERVENTIONS:
Diagnostic Test: MIBI scintigraphy — Performing a MIBI scintigraphy, then, in the case of negativity, a single F18-choline PET
  Other Names: F18-choline PET
Diagnostic Test: F18-choline PET — Realization of a F18-choline PET, then, in case of negativity, a MIBI scintigraphy
  Other Names: MIBI scintigraphy

SUMMARY:
The investigators hypothesize that positron emission tomography with fluorocholline (F18-choline PET) will reduce the proportion of unnecessary invasive surgery decisions and that the higher cost of positron emission tomography versus MIBI scintigraphy (Tc99m-sestaMIBI ) will be offset by lower cost in terms of type. surgery performed wisely and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old
* Patient presenting with primary hyperparathyroidism and for whom an excisional surgery is planned
* For women of childbearing age, negative pregnancy test at Baseline
* Biological assessment confirming the diagnosis of primary hyperparathyroidism (high serum PTH and calcium concentrations)
* Affiliation to a social security scheme
* Patient having signed his written consent

Exclusion Criteria:

* Patient deprived of liberty, under tutorship or curatorship
* Hypersensitivity to TECNESCAN SESTAMIBI
* Any associated medical or psychological condition that could compromise the patient's ability to participate in the study
* Pregnant or lactating woman
* History of parathyroid surgery
* Patient with multiple endocrine neoplasia 1 (NEM1)
* Known hypersensitivity to fluorocholine or to any of the excipients (sodium chloride, water for injections)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Compare, between each diagnostic strategy, the proportion of patients for whom the first-line imaging technique guided the surgical procedure wisely | Up to 2 months

SECONDARY OUTCOMES:
Estimate the diagnostic performance of each strategy by measuring sensitivity and specificity | Up to 2 months
Evaluate post-surgical complications by measuring tne number of infections, hematoma | Up to 2 months

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Brest, Brest
  - Centre François Baclesse, Caen
  - Centre Eugène Marquis, Rennes
  - CHU, Rennes

REFERENCES:
- [Derived] Quak E, Lasne-Cardon A, Cavarec M, Lireux B, Bastit V, Roudaut N, Salaun PY, Keromnes N, Potard G, Vaduva P, Esvant A, Jegoux F, de Crouy-Chanel O, Devillers A, Guery C, Lasnon C, Ciappuccini R, Legrand B, Estienne A, Christy F, Grellard JM, Bardet S, Clarisse B. F18-Choline PET/CT or MIBI SPECT/CT in the Surgical Management of Primary Hyperparathyroidism: A Diagnostic Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Aug 1;150(8):658-665. doi: 10.1001/jamaoto.2024.1421. PMID 38900416
- [Derived] Quak E, Lasne Cardon A, Ciappuccini R, Lasnon C, Bastit V, Le Henaff V, Lireux B, Foucras G, Jaudet C, Berchi C, Grellard JM, Lequesne J, Clarisse B, Bardet S. Upfront F18-choline PET/CT versus Tc99m-sestaMIBI SPECT/CT guided surgery in primary hyperparathyroidism: the randomized phase III diagnostic trial APACH2. BMC Endocr Disord. 2021 Jan 7;21(1):3. doi: 10.1186/s12902-020-00667-5. PMID 33413316